CLINICAL TRIAL: NCT02414048
Title: Predictive Methods Determining Tumour Hypoxia in Head and Neck Cancer Patients - a Prospective Project
Brief Title: Hypoxia Analysis in Head and/or Neck Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marius Gustav Bredell (Other)
Responsible Party: Sponsor-Investigator, Marius Gustav Bredell, Dr, University of Zurich
Organization: University of Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KEK-Nr.2014-0393
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Head and Neck Cancer
Keywords: Hypoxia; Head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Hypoxia | interventions — pimonidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pimonidazole (Other): All patients will receive Pimonidazole to demarcate hypoxia regions in the tumour
  Interventions: Drug: Pimonidazole

INTERVENTIONS:
Drug: Pimonidazole — Pimonidazole will be administered orally and will serve to demarcate the hypoxic areas in the tumour
  Other Names: Oral Hypoxyprobe

SUMMARY:
The primary objective is the prospective determination of disease-specific and overall survival in head and neck cancer patients who have undergone surgery, correlated to non-invasive methods of measuring tumour hypoxia.

The secondary objective is to define tumour hypoxia using non-invasive methodology.

DETAILED DESCRIPTION:
The incidence of head and neck squamous cell cancer (HNSCC) is around 600 000 cases per year worldwide. The main sites for HNSCC are the larynx, the pharynx and the oral cavity. Head and neck cancers, however, also include salivary gland tumours, as well as nasopharyngeal cancer and paranasal and nasal sinus cancer but these are rare. The major risk factors are smoking, alcohol abuse and Human Papillomavirus (HPV) infection. In spite of radical surgical treatment and aggressive neo-adjuvant and adjuvant therapies, the prognosis of head and neck cancer is very poor due to the fact that the tumours are often hypoxic.

Tumour hypoxia is heterogenous and results from an imbalance between oxygen supply and oxygen consumption. Acute hypoxia is caused by abnormal structure and function of the microvasculature supplying the tumour. Chronic hypoxia is caused by the increased distance through which the oxygen has to diffuse to get from the blood vessels to the tumour cells and by the reduced oxygen caused by the anaemia which can be treatment or disease-related. These hypoxic regions have been shown to affect the metabolism of the cells, making them more aggressive with increased risk of metastasis and a worse prognosis. Also, because radiotherapy relies on oxygen to cause maximal cytotoxicity, a lack of oxygen to the cells or even a lack of oxygen consumption by the cells would cause a decrease in the effectiveness of the radiotherapy and the cytotoxicity. Hypoxic cells have an acidic environment which affects drug delivery and drug activity, so chemotherapy is compromised.

In order to predict outcome and identify patients with a worse prognosis or patients that would benefit from appropriate treatments, in vivo measurement of tumour hypoxia is required. Numerous methods have been explored but there is no accepted gold standard. Imaging and biomarker analysis have been shown to have potential but the data are insufficient. In this project the investigators would prospectively use existing imaging techniques and analysis of various bodily fluids to predict outcome. This is a collaboration between 5 different departments so that as much information as possible can be analysed and used to come to a possible solution.

ELIGIBILITY:
Inclusion Criteria:

* Malignancy in head and/or neck region only
* Interdisciplinary Head and neck tumour board (USZ) confirmed inclusion in the project
* For patients with reproductive potential (e.g. female participants who are surgically sterilised/hysterectomised or post-menopausal for longer than 2 years are not considered as beig of child bearing potential), a willingness to use adequate contraceptive measures to prevent pregnancy during the project.

Exclusion Criteria:

* Pregnant or breastfeeding
* Suffers from claustrophobia
* Known allergy to Pimonidazole
* Participation in a study with an investigational drug within the 30 days preceding and during this project
* Tumour size smaller than 1cm
* Has symptomatic Chronic Obstructive Pulmonary Disease (COPD)
* Patient refuses or is unable to give a written informed consent
* Previous treatment for head and/or neck cancer
* Inability to follow the procedures of the project e.g. due to language problems, psychological disorders, dementia, etc. of the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-04; Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Disease-specific and overall survival correlated with tumour hypoxia | 5-years
  Tumour hypoxia will be determined from the Pimonidazole staining and this will be correlated to disease-specific survival and overall survival. The study has been approved for 10 participants to be increased by the ethical committee to 100 once the study is going.

CONTACTS AND LOCATIONS:
Overall Officials: Marius Bredell, Principal Investigator — Department of Cranio-, Maxillofacial and Oral Surgery, University Hospital Zurich
Locations (1):
- Department of Cranio-, Maxillofacial and Oral Surgery, Zurich, Switzerland